CLINICAL TRIAL: NCT01046604
Title: Mitigating Cardiac Inflammation and Oxidative Stress in Atrial Myocardium Via Short-term Lovaza Treatment Prior to Surgery
Brief Title: Pilot Study of Lovaza (Omega 3 Fatty Acids) to Improve Cardiac Antioxidant/Anti-inflammatory Profile Before Cardiac Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: East Carolina University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Ethan J. Anderson, Assistant Professor, East Carolina University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ECUomega3-01
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-08

CONDITIONS: Mitral Valve Regurgitation; Left Atrium Dilatation and Hypertrophy; Mitochondrial Dysfunction in the Heart; Cardiomyocyte Apoptosis; Cardiac Inflammation
Keywords: mitral valve regurgitation; omega 3 fatty acids; fish oil; cardiac; mitochondria; apoptosis; human heart
MeSH Terms: conditions — Mitral Valve Insufficiency; Hypertrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No treatment (No Intervention): This is the group of patients that will not undergo any treatment with Lovaza prior to mitral valve repair surgery. This is the 'control' group.
- Lovaza treated (Active Comparator): This arm will be the group of patients that will be treated with Lovaza prior to undergoing mitral valve repair surgery.
  Interventions: Drug: Lovaza group

INTERVENTIONS:
Drug: Lovaza group — Patients who are scheduled for mitral valve repair surgery at least 3 weeks removed from the initial consult will be recruited to take 4 capsules of Lovaza (omega 3 fatty acids) daily, for 3 weeks prior to their surgery.
  Other Names: omega 3 fatty acid esters
  Arms: Lovaza treated

SUMMARY:
In the absence of treatment, severe mitral valve regurgitation (MR) results in left atrium (LA) dilatation and hypertrophy, followed ultimately by left ventricular dysfunction and heart failure. One promising intervention for the prevention of the deleterious effects of pressure overload-induced cardiac hypertrophy and heart failure is dietary supplementation with n-3 polyunsaturated fatty acids (PUFAs). However, the molecular targets and mechanisms by which n-3 PUFAs exert their effects are not completely defined. A possible target of n-3 PUFAs is the mitochondrial membrane which has broad implications given that mitochondrial dysfunction and altered metabolism have been associated with cardiac hypertrophy and heart failure. The investigators have recently identified significant mitochondrial dysfunction in the LA of patients with severe MR, as compared to their non-hypertrophied right atrium (RA). However, the investigators have not addressed the possibility that intervention with purified n-3 PUFAs (Lovaza) could improve mitochondrial function. From a mechanistic perspective, the investigators have observed in vitro that n-3 PUFAs accumulate predominately into the mitochondrial membrane of cardiomyocytes where the investigators believe they exert their effects on the biophysical organization of the membrane. Therefore, the CENTRAL HYPOTHESIS is that administering Lovaza to patients with severe MR will reduce apoptosis and improve mitochondrial function in LA (Aim 1). This change in mitochondrial function will be driven by significant biochemical and biophysical remodeling of the mitochondrial membrane (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18+ undergoing minimally invasive mitral valve repair surgery will be enrolled in this study.

Exclusion Criteria:

* Patients with chronic renal insufficiency
* Chronic obstructive pulmonary disease
* Previous myocardial infarction
* Left ventricular dysfunction (ejection fraction <40%)
* Use of anti-arrhythmic drugs other than beta blockers, and the presence of an implantable defibrillator.
* In addition, patients that have a high dietary intake of fish (≥ 2 servings/week) or have been taking n-3 PUFA supplements will be excluded.
* Also, patients that are allergic to fish or shellfish, or taking any anticoagulant/antiplatelet medications other than aspirin (e.g. Plavix, Coumadin) will be excluded from this study.
* Patients under the age of 18, and women who are pregnant will be excluded from this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Specific Aim 1: To determine if Lovaza treatment reduces markers of inflammation and improves mitochondrial function in atrial myocardium | 15 months

SECONDARY OUTCOMES:
Specific Aim 2: To determine if Lovaza treatment alters the biophysical and biochemical organization of cardiac mitochondrial membranes. The following questions will be addressed using the blood and cardiac tissue samples collected as described above: | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Ethan J Anderson, PhD, Principal Investigator — Assistant Professor, Department of Pharmacology and Toxicology, East Carolina University
Locations (1):
- Brody School of Medicine, Greenville, North Carolina, United States